CLINICAL TRIAL: NCT07229703
Title: Burst Abdomen Surgery
Brief Title: Management of Burst Abdomen
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Tamer.A.A.M.Habeeb, prof, Zagazig University
Other Study IDs: burst abdomen management
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Burst Abdomen
Keywords: tension suture; burst abdomen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- component separation: management of burst abdomen by component separation
  Interventions: Procedure: component separation
- primary repair: primary repair of burst abdomen
  Interventions: Procedure: primary repair for burst abdomen

INTERVENTIONS:
Procedure: component separation — component separation for management of burst abdomen
  Groups: component separation
Procedure: primary repair for burst abdomen — management of burst abdomen by primary repair
  Groups: primary repair

SUMMARY:
The goal of this observational study is to learn about the long-term effects of repair of burst abdomen by both primary repair and component separation. The main question it aims to answer is:

Does component separation lower postoperative complications ?

DETAILED DESCRIPTION:
to compare between 2 common techniques for management of burst abdomen

ELIGIBILITY:
Inclusion Criteria:

* adult patients (≥18 years) underwent PCS+TAR+MA or primary suture with tension sutures for complete burst abdomen

Exclusion Criteria:

* 1. BA grade 1B, 2, 3, and 4 (n=17),
* < 18 years (n=2)
* Primary laparotomy performed through a non-midline incision (n=4)
* Open abdomen (n=5)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: > 18 years with BA
Sampling Method: Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
wound infection | 30 days

SECONDARY OUTCOMES:
incisional hernia | 5 years

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: Related Info — http://tameralnaimy@hotmail.com